CLINICAL TRIAL: NCT02136927
Title: Bioavailability Study of SPARC1210 and Reference1210 in Subjects With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLR_12_10
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPARC1210 (Experimental): Intravenous administration of SPARC1210
  Interventions: Drug: SPARC1210
- Reference1210 (Active Comparator): Intravenous administration of Reference1210
  Interventions: Drug: Reference1210

INTERVENTIONS:
Drug: SPARC1210
  Arms: SPARC1210
Drug: Reference1210
  Arms: Reference1210

SUMMARY:
Pharmacokinetic, bioequivalence study

ELIGIBILITY:
Inclusion Criteria:

* The subject has given written, informed consent and is available for the entire study.
* Histologically or cytologically confirmed diagnosis of breast cancer;
* Locally recurrent or metastatic breast cancer for which taxane-based therapy is a rational treatment option;
* Age 18 years or more

Exclusion Criteria:

* Known hypersensitivity to both the study drugs or its excipients (Cholesteryl sulfate, Caprylic acid, Polyvinylpyrrolidone, Ethanol or Polyethylene glycol);
* Presence of clinically evident active CNS metastases, including leptomeningial involvement, requiring steroid or radiation therapy;
* Pre-existing clinically significant peripheral neuropathy (Grade 2 or higher according to CTCAE, Version 4.0);
* Any other severe concurrent disease which in the judgment of the investigator would make the subject inappropriate for entry into this study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Pre-dose, post-dose up to 3 days
  Samples will be collected from all subjects at scheduled time-points: pre-dose and up to 3 days post-dose.

OTHER OUTCOMES:
Adverse events | Day 3
  AEs encountered following dosing with PICN or Abraxane® will be recorded as per CTCAE, Version 4.0

CONTACTS AND LOCATIONS:
Locations (12):
- India (12):
  - SPARC Site 12, Hyderabad, Andhra Pradesh
  - SPARC Site 9, Hyderabad, Andhra Pradesh
  - SPARC Site 2, Goraj, Gujarat
  - SPARC Site 8, Kochi, Kerala
  - SPARC Site 11, Mumbai, Maharashtra
  - SPARC Site 5, Nagpur, Maharashtra
  - SPARC Site 4, Nashik, Maharashtra
  - SPARC Site 1, Pune, Maharashtra
  - SPARC Site 3, Pune, Maharashtra
  - SPARC Site 6, New Delhi, National Capital Territory of Delhi
  - SPARC Site 10, Chennai, Tamil Nadu
  - SPARC Site 7, Madurai, Tamil Nadu